CLINICAL TRIAL: NCT01338844
Title: A Prospective, Randomized, Double Blind, Study on the Clinical Efficacy Myo-inositol Versus D-chiro-inositol in Women Undergoing in Vitro Fertilization Embryo Transfer.
Brief Title: Role of Myo-inositol and D-chiro-inositol on Oocyte Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Collaborators: Research Center for Reproductive Medicine Villa Mafalda (Unknown); San Raffaele University Hospital, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MI_vs_DCI_Oo_q
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-04

CONDITIONS: Infertility
Keywords: Poor oocyte quality; IVF failure
MeSH Terms: conditions — Infertility | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-Chiro-inositol (Experimental): Patients will receive 1.2g/day of D-chiro-inositol
  Interventions: Dietary Supplement: D-chito-Inositol
- Myo-inositol (Active Comparator): Patients will receive 4g/day of myo-inositol
  Interventions: Dietary Supplement: Myo-inositol

INTERVENTIONS:
Dietary Supplement: Myo-inositol
  Arms: Myo-inositol
Dietary Supplement: D-chito-Inositol
  Arms: D-Chiro-inositol

SUMMARY:
Controlled ovarian hyperstimulation with gonadotropins is an integral part of the various stimulation protocols for patients undergoing in-vitro fertilization (IVF) and other Assisted Reproductive Technologies (ART) such as intracytoplasmic sperm injection (ICSI).

The hormonal control of multiple follicular growth and maturation is a critical part of ART procedures since it maximizes the yield of embryos to be transferred, thus increasing the cumulative pregnancy rate.

Recent studies have shown the efficacy of myo-inositol (MI) supplementation as a simple and highly effective treatment in order to improve oocyte quality in patients undergoing IVF. Indeed, it was previously shown that MI follicular fluid (FF) concentration is a reliable predictor of oocyte quality. High MI concentration in the FF directly correlates with high oocyte and embryo quality.

Another stereoisomer of Inositol was successfully used into clinical practice D-chiro-inositol (DCI). In particular, DCI supplementation was used to restore ovulation in hyperglycemic PCOS patients.

In the present study we aim to compare MI versus DCI supplementation on oocyte quality of women undergoing IVF-ET

ELIGIBILITY:
Inclusion Criteria:

* women undergoing IVF treatments
* Body mass index <28
* FSH <10IU/L
* Normal uterine cavity, anatomy and functions

Exclusion Criteria:

* PCOS
* Stage III or IV endometriosis
* Premature ovarian failure
* Poor responder

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
number of morphologically mature oocytes
Total international units (IU) of recombinant FSH administrated
number of grade 1 embryos

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Carlomagno, Ph.D., Principal Investigator — AGUNCO Obstetrics and Gynecology Centre; Vittorio Unfer, M.D., Principal Investigator — AGUNCO Obstetrics and Gynecology Centre; Franco Lisi, M.D., Principal Investigator — Research Center for Reproductive Medicine; Enrico Papaleo, M.D., Principal Investigator — San Raffaele Hospital; Scott Roseff, MD, Principal Investigator — The Palm Beach Center for Reproductive Medicine
Locations (3):
- Italy (3):
  - San Raffaele Hospital, Milan
  - Research Center for Reproductive Medicine Villa Mafalda, Roma
  - Agunco, Rome

REFERENCES:
- [Background] Chiu TT, Rogers MS, Law EL, Briton-Jones CM, Cheung LP, Haines CJ. Follicular fluid and serum concentrations of myo-inositol in patients undergoing IVF: relationship with oocyte quality. Hum Reprod. 2002 Jun;17(6):1591-6. doi: 10.1093/humrep/17.6.1591. PMID 12042283
- [Background] Unfer V, Raffone E, Rizzo P, Buffo S. Effect of a supplementation with myo-inositol plus melatonin on oocyte quality in women who failed to conceive in previous in vitro fertilization cycles for poor oocyte quality: a prospective, longitudinal, cohort study. Gynecol Endocrinol. 2011 Nov;27(11):857-61. doi: 10.3109/09513590.2011.564687. Epub 2011 Apr 5. PMID 21463230
- [Background] Rizzo P, Raffone E, Benedetto V. Effect of the treatment with myo-inositol plus folic acid plus melatonin in comparison with a treatment with myo-inositol plus folic acid on oocyte quality and pregnancy outcome in IVF cycles. A prospective, clinical trial. Eur Rev Med Pharmacol Sci. 2010 Jun;14(6):555-61. PMID 20712264
- [Background] Papaleo E, Unfer V, Baillargeon JP, Chiu TT. Contribution of myo-inositol to reproduction. Eur J Obstet Gynecol Reprod Biol. 2009 Dec;147(2):120-3. doi: 10.1016/j.ejogrb.2009.09.008. Epub 2009 Oct 2. PMID 19800728
- [Background] Papaleo E, Unfer V, Baillargeon JP, Fusi F, Occhi F, De Santis L. RETRACTED: Myo-inositol may improve oocyte quality in intracytoplasmic sperm injection cycles. A prospective, controlled, randomized trial. Fertil Steril. 2009 May;91(5):1750-1754. doi: 10.1016/j.fertnstert.2008.01.088. Epub 2008 May 7. PMID 18462730
- [Background] Nestler JE, Jakubowicz DJ, Reamer P, Gunn RD, Allan G. Ovulatory and metabolic effects of D-chiro-inositol in the polycystic ovary syndrome. N Engl J Med. 1999 Apr 29;340(17):1314-20. doi: 10.1056/NEJM199904293401703. PMID 10219066